CLINICAL TRIAL: NCT07117422
Title: Efficacy and Safety of Venetoclax Plus Decitabine in Elderly/Unfit Patients With Newly Diagnosed AML: A Multicenter Single-Arm Study
Brief Title: Venetoclax-Decitabine in Untreated Elderly/Unfit AML
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Hebei Medical University (Other)
Collaborators: Handan First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-R010-F1
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VEN+DEC (Experimental)
  Interventions: Drug: VEN + DEC

INTERVENTIONS:
Drug: VEN + DEC — Induction regimen
  Venetoclax (VEN): Day1-10
  Decitabine (DEC):20mg/m²/day, Day 2-4
  20mg/m² every 8 hours, Day 5-6
  FLT3 Inhibitors (for FLT3/ITD+ patients only):
  Sorafenib or Gilteritinib, Day 8-14
  Post-Remission Treatment
  Venetoclax (VEN): 400 mg/day, Day 1-7
  Decitabine (DEC): 20 mg/m² every 8 hours, Day 2-3 (Regimen repeated every 4-6 weeks)
  FLT3 Inhibitors (for FLT3/ITD+ patients only):
  Sorafenib or Gilteritinib, Day 8-14

SUMMARY:
Acute myeloid leukemia (AML) is a highly fatal malignancy in China, with particularly poor outcomes in elderly patients. Low-intensity regimens yield low remission rates, and median overall survival (OS) typically remains under 6-9 months. Venetoclax (VEN) combined with hypomethylating agents (azacitidine or decitabine（DEC）) has emerged as a first-line therapy for these patients, significantly improving response rates and survival. However, challenges persist, including suboptimal complete remission (CR) rates, low Measurable Residual Disease（MRD） negativity, and tolerability issues with prolonged use.

Recent studies suggest that a 3-day decitabine regimen combined with VEN may enhance efficacy and tolerability. Building on prior evidence and our institutional experience, we propose this study to evaluate an optimized dosing strategy of VEN plus decitabine in treatment-naïve elderly or chemotherapy-ineligible AML patients, aiming to further improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting the World Health Organization (WHO) 2022 diagnostic criteria for acute myeloid leukemia (AML), excluding:Acute promyelocytic leukemia (APL)

   AML with recurrent genetic abnormalities, including:t(8;21)(RUNX1::RUNX1T1)

   inv(16)(p13.1q22) or t(16;16)(p13.1q22)/CBFβ::MYH11
2. Patients classified as AML, not otherwise specified (NOS) per WHO criteria, excluding:Acute panmyelosis with myelofibrosis 、Myeloid sarcoma
3. Age and fitness criteria:

   -Group A: Age ≥65 years (unwilling to receive intensive chemotherapy)

   Group B: Age >18 years and ineligible for standard-dose chemotherapy, defined by ≥1 of the following:ECOG performance status 2 or 3；History of chronic heart failure (CHF) requiring treatment or left ventricular ejection fraction (LVEF) ≤50% DLCO ≤65% or FEV1 ≤65%Creatinine clearance ≥30 mL/min but ≤45 mL/min (Cockcroft-Gault or 24-hour urine collection)、Any other condition deemed incompatible with standard chemotherapy (requires PI approval)
4. No prior AML therapy, except:Hydroxyurea、Low-dose cytarabine (<1.0 g/day)
5. ECOG performance status ≤3
6. Laboratory requirements (within 7 days prior to treatment):AST/ALT/ALP ≤3×ULN (≤5×ULN if due to leukemic involvement)、Total bilirubin ≤2×ULN、Cardiac enzymes <2×ULN、Serum creatinine clearance ≥30 mL/min (measured or calculated)
7. Contraception requirements:Negative pregnancy test (within 72 hours before treatment) for women of childbearing potential；Agreement to use effective contraception during treatment and for 3 years after therapy
8. Life expectancy ≥2 months
9. Informed consent:Signed by patient, legal guardian, or immediate family member (if patient is unable to consent due to medical condition)

Exclusion Criteria:

1. AML with BCR::ABL1 fusion or chronic myeloid leukemia (CML) in blast crisis.
2. Previously treated AML patients (received prior induction chemotherapy, regardless of response).
3. Secondary AML, including:Therapy-related AML (per WHO classification)、AML with prior history of myelodysplastic syndrome (MDS) or myeloproliferative neoplasm (MPN)
4. Concurrent hematologic disorders (e.g., hemophilia, myelofibrosis, or other conditions deemed ineligible by the investigator). Exception: Patients with prior blood count abnormalities but confirmed non-MDS/MPN by bone marrow examination may be included.
5. Pregnant or lactating women.
6. Hypersensitivity to any study drugs.
7. Use of strong/moderate CYP3A4 inducers within 3 days prior to treatment initiation.
8. Active malignancy in other organs (requiring treatment).
9. Clinically significant hepatic/renal dysfunction exceeding inclusion criteria limits.
10. Active cardiac disease, defined as ≥1 of the following:Myocardial infarction within 6 months before enrollment；History of symptomatic arrhythmia requiring medication；Uncontrolled/symptomatic congestive heart failure (NYHA Class >2)
11. Active infections, including:Untreated tuberculosis or pulmonary aspergillosis

    Known HIV, active hepatitis B (HBV), or hepatitis C (HCV)
12. Central nervous system (CNS) leukemia at baseline.
13. Medical history of:Epilepsy requiring medication、Dementia or psychiatric disorders impairing protocol compliance
14. Conditions limiting oral drug absorption (e.g., malabsorption syndrome).
15. Investigator's discretion for ineligibility.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
the Complete Remission (CR) Rate after Cycle 1 | up to 42 days after treatment

SECONDARY OUTCOMES:
Overall Survival (OS) | Within 5 years after randomization
Relapse-Free Survival Rate (RFS) | Within 5 years after randomization
Cumulative incidence of relapse | Within 5 years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: LING XI GUO, Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- The Second Hospital of Hebei Medical University, Hebei, China

IPD SHARING:
Plan to Share IPD: No